CLINICAL TRIAL: NCT03247660
Title: Effectiveness of the Perineal Physiotherapy in the Prevention and Treatment of Pelvic Floor Dysfunction in Postpartum
Brief Title: Perineal Physiotherapy in Postpartum
Acronym: PT-POSTPARTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21/2013
Record Dates: First submitted 2017-08-05; First posted 2017-08-14 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Post Partum

STUDY DESIGN:
Intervention Model Description: 3 groups: 2 experimental groups and 1 control group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PFMT&HE group (Experimental): A directly pelvic floor muscle (PFM) training protocol will be applied. Participants will performed PFM exercises in the way proposed by the PERFECT scheme. Biofeedback exercises will be also performed in lithotomy position. If the evolution of the women will allow it, the last two treatment biofeedback sessions will be conducted in standing position, to train PFM in more challenging and functional situation. In this group participants will be also trained hypopressive breathing and will perform five hypopressive exercises: two postures in supine, one on four-kneeling, and two in standing position. Educational strategy will also be applied. The intervention will last 8 weeks, 2 sessions per week. Each session will last 40/50 minutes.
  Interventions: Other: PFM training; Other: HE; Behavioral: Educational strategy
- HE group (Experimental): Women will be instructed in thirty-three Hypopressives exercises (HE) described by the developer of the Hypopressive Abdominal Gymnastics, Dr. Caufriez plus Educational strategy.
  The intervention will last 8 weeks, 2 sessions per week. Each session will last 40/50 minutes.
  Interventions: Other: HE; Behavioral: Educational strategy
- Control group (Active Comparator): The educational strategy will consist of instruction of printed materials and dimensional anatomical models about the anatomy of the pelvic floor and the physiology of the pelvic organs. It will be recommended to avoid risk factors, such as gaining weight, weight lifting, high impact sports, constipation, smoking, or drinking too much caffeine. They will also instruct in toilet habits, and will be taught to use the knack maneuver before and during increases of intra-abdominal pressure. The intervention will last 8 weeks, 1 session per week. Each session will last 40/50 minutes.
  Interventions: Behavioral: Educational strategy

INTERVENTIONS:
Other: PFM training — See information included in arm/group descriptions.
  Other Names: Pelvic floor muscle training
  Arms: PFMT&HE group
Other: HE — See information included in arm/group descriptions.
  Other Names: Hypopressive exercises
  Arms: HE group; PFMT&HE group
Behavioral: Educational strategy — See information included in arm/group descriptions.

SUMMARY:
Objective: To find out the effectiveness of pelvic-perineal physiotherapy in prevention and treatment of postpartum pelvic floor dysfunction caused by vaginal delivery.

DETAILED DESCRIPTION:
Design: Randomized, controlled and single blinded clinical trial. Participants will be randomly assigned to one of these groups: Experimental group: pelvic-perineal physical therapy plus hypopressive exercises plus training in lifestyle advice; Experimental group II: hypopressive exercises plus training in lifestyle advice; Control group: just training in lifestyle advice. In the 3 groups several physical therapy assessments will be undertaken: 1st before intervention, 2nd immediately after completing intervention; 3th, 4th, 5th and 6th after 3, 6, 12 and 24 months. Study subjects: Postnatal women (6 and 8 weeks after vaginal delivery), primiparous, whose vaginal delivery has occurred in the "PrÍncipe de Asturias" Hospital, which have not been already treated for pelvic floor dysfunction, and after reading, understanding and freely signing an informed consent form. Sample size: 240 subjects will be included (80 subjects per group). Allowing for 15% of drop-outs and taking into account that 17% of women in the intervention group may develop pelvic floor dysfunction (urinary incontinence) versus 40% in the control group, with an alpha risk of 0.05, a beta risk of 0.1 in a bilateral contrast using the arcsine approximation. Data analysis: A descriptive analysis will be done of all variables. A confidence level of 95% (p <0,05) will be established for all the cases. Effectiveness will be evaluated by comparing between the two groups of the change in outcome variables between visits.

ELIGIBILITY:
Inclusion Criteria:

* Postnatal women (6 and 8 weeks after vaginal delivery)
* Primiparous
* Whose vaginal delivery has occurred in the "Príncipe de Asturias" Hospital
* Women have not been already treated for pelvic floor dysfunction
* Women reading, understanding and freely signing an informed consent form

Exclusion Criteria:

* Postnatal women with medical diagnosis of pelvic floor dysfunction (PFD) prior to pregnancy and delivery
* Women with a history of conservative treatment or PFD surgery
* Women with concomitant or systemic disease that may affect the treatment (neurological, gynecological, urological or connective tissue), or with active or recurrent urinary infection without treatment at the time of the intervention proposed in this study, or hematuria
* Postnatal women with cognitive limitations to understand information, respond to questionnaires, consent and / or participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Change in life impact of pelvic floor dysfunction | 5 assessments to evaluate change from baseline: at baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be assessed by the PFIQ-7 Spanish version. The PFIQ-7 consists of 3 scales of 7 questions each taken from the Urinary Impact Questionnaire, the Pelvic Organ Prolapse Impact Questionnaire, and the Colorectal-Anal Impact Questionnaire. The 3 scales are scored from 0 (least impact) to 100 (greatest impact) and an overall summary score (0 to 300).
Change in symptoms and quality of life | 5 assessments to evaluate change from baseline: at baseline, after the intervention period (2 months from baseline), , 3 months, 6 months and 12 months after the intervention.
  It will be assessed by PFDI-20 that is both a symptom inventory and a measure of the degree of bother and distress caused by pelvic floor symptoms. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300 and the higher the score, the worse quality of life. The 3 scales include questions taken from the following widely used outcome measures: Urinary Distress Inventory - 6 questions, Pelvic Organ Prolapse Distress Inventory - 6 questions, and Colorectal-Anal Distress Inventory - 8 questions collecting data about UI, POP and colorectal and anal symptoms.
Change in pelvic floor muscle strength | 5 assessments to evaluate change from baseline: at baseline, after the intervention period (2 months from baseline), , 3 months, 6 months and 12 months after the intervention.
  It will be measured with manometry (cm2O2)
Change in pelvic floor muscle characteristics | 5 assessments to evaluate change from baseline: at baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  Vaginal palpation will qualify PFM condition using the Levator any test (LAT) ranging from 0 to 5, according to the muscles strength and endurance.
Change in pelvic floor muscle strength | 5 assessments to evaluate change from baseline: at baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be measured with dynamometry (gr)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alcalá. FPSM research group. HUPA, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735